CLINICAL TRIAL: NCT03605732
Title: The Effectiveness of an Educational Intervention Based on Self-help for Sleep Hygiene Promotion on Employees of Qazvin University of Medical Sciences
Brief Title: The Effectiveness of an Educational Intervention Based on Self-help for Sleep Hygiene Promotion on Patients With Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir H Pakpour, Supervisor, Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IR.QUMS.REC.1396.455
Record Dates: First submitted 2018-07-22; First posted 2018-07-30 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Insomnia; Behavioral Intervention
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Intervention group: They will receive an educational app designed to improve sleep, and will receive self-help training in a six-week training package.
  Interventions: Behavioral: self help sleep hygiene intervention application
- Patient education (Active Comparator): Patients will receive written weekly information on accurate and relevant information regarding insomnia symptoms, physiological controls of sleep, sleep hygiene practices, healthy sleep behaviors
  Interventions: Other: patients education

INTERVENTIONS:
Behavioral: self help sleep hygiene intervention application — This intervention lasts for six weeks. The intervention is App-based and mainly consists of the most potent CBT techniques as well Health action process approach. Weekly feedback is provided by health psychologists.
  Arms: intervention
Other: patients education — Participants in the PE group will receive written weekly information on accurate and relevant information regarding insomnia symptoms, physiological controls of sleep, sleep hygiene practices, healthy sleep behaviors
  Arms: Patient education

SUMMARY:
This plan will be implemented on the staff of the Qazvin University of Medical Sciences. The Insomnia Severity Index questionnaire will be used to screen for insomnia and low sleep health. This questionnaire is provided online to the staff through communication channels such as telegrams to help people who are interested in participating in this research. Individuals who scored more than 8 were randomly assigned to intervention and control groups and completed the Insomnia Index Index. The intervention group will then receive an app-based educational intervention designed to improve sleep hygiene. Control group: Participants in the control group perform routine activities. The intervention and control group will fill out the relevant questionnaire one and three and six months after the completion of the training to assess the impact of the intervention online.

ELIGIBILITY:
Inclusion Criteria:

* Clinical level of Insomnia (more than 10 on ISI)
* Meets criteria for Insomnia according to DSM-IV-TR
* Enough language skills
* Have access to an Android smartphone or a desktop computer with Internet access
* Participants will be required to sign an informed consent form

Exclusion Criteria:

* Uncontrolled medical condition suspected to interfere with sleep or requiring immediate treatment outside of the study
* Alcohol/drugs abuse
* Participation in other trials concurrently
* pregnancy
* having children under 2 years old
* Not having an internet-connected computer, cellular phone or tablet
* Working night shifts
* Somatic or psychiatric conditions requiring acute care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-04-06 (Actual); Study Completion 2019-06-08 (Actual)

PRIMARY OUTCOMES:
Sleep Quality | changes in PSQI baseline , 1 month, 3 months and 6 months follow-up
  The Pittsburgh Sleep Quality Index includes seven components of subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, the use of sleep medications and day time dysfunctions provide a total score of these seven components that allows us to better understand the quality and quantity of one's sleep. The Pittsburgh Sleep Quality Index is a self-reporting instrument consisting of nine questions designed to measure the quality of sleep disorders in a period of one month. The scale scores range from 0 to 21, with higher scores indicating poor quality of sleep and scores less than 5 considered as high quality of sleep
sleep hygiene behavior | changes in sleep hygiene behavior baseline , 1 month, 3 months and 6 months follow-up
  Sleep hygiene behaviour will use three items to measure how many days the participants had good sleep hygiene.
  behaviour.

SECONDARY OUTCOMES:
Anxiety and Depression | changes in Anxiety and Depression baseline , 1 month, 3 months and 6 months follow-up
  Zigmond and Snaith developed the 14-item HADS to measure the anxiety (7 items) and depression (7 items) of patients with both somatic and mental problems. The response descriptors of all items are Yes, definitely (score 3); Yes, sometimes (score 2); No, not much (score 1); No, not at all (score 0); except for items 7 and 10, which are scored reversely. A higher score represents higher levels of anxiety and depression: a domain score of 11 or greater indicates anxiety or depression; 8-10 indicates borderline case; 7 or lower indicates no signs of anxiety or depression. The two-factor framework of the HADS has been supported in cancer patients.
Psychological predictors of sleep hygiene behavior (intention, planning, outcome expectancies,Habit,Self-monitoring,Self-efficacy) | changes from baseline , changes from baseline , 1 month and 6 Months follow-up
  psychological predictors of sleep hygiene behavior will be assessed using a using a self-reported measure. All items are rated on a Likert-type scale, ranging from 1 to 5.

CONTACTS AND LOCATIONS:
Locations (1):
- Qazvin University of Medical Sciences, Qazvin, Iran

REFERENCES:
- [Derived] Rajabi Majd N, Brostrom A, Ulander M, Lin CY, Griffiths MD, Imani V, Ahorsu DK, Ohayon MM, Pakpour AH. Efficacy of a Theory-Based Cognitive Behavioral Technique App-Based Intervention for Patients With Insomnia: Randomized Controlled Trial. J Med Internet Res. 2020 Apr 1;22(4):e15841. doi: 10.2196/15841. PMID 32234700